CLINICAL TRIAL: NCT00127140
Title: A Phase I Clinical Study of MK0683 in Patients With Malignant Lymphoma
Brief Title: A Study of Oral Suberoylanilide Hydroxamic Acid (SAHA) in Patients With Malignant Lymphoma (0683-030)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0683-030; 2005_041
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vorinostat (Experimental): Participants received (Cycle 1) once-daily vorinostat at assigned dose (100 or 200 mg) on Days 1 and 17 and twice-daily on Days 3-16. Thereafter, participants remaining on study received the same dose level therapy twice-daily for 14 consecutive days followed by 7 days of rest.
  Interventions: Drug: vorinostat

INTERVENTIONS:
Drug: vorinostat

SUMMARY:
The primary purpose of this trial is to determine the maximum tolerated dose (MTD), or the maximum acceptable dose (MAD) and evaluate the dose limiting toxicity (DLT) of oral vorinostat in patients with malignant lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients who relapsed after complete or partial response, or ineffective in previous chemotherapy

Exclusion Criteria:

* Patients with history of chemotherapy, antibody therapy, radiotherapy, during the previous 4 weeks (6 months for radioisotope-labeled antibody)
* Any uncontrolled concomitant illness
* Are pregnant or breast-feeding
* Serious drug or food allergy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Number of participants Experiencing Dose-Limiting Toxicities (DLTs) | Up to 21 days

SECONDARY OUTCOMES:
Area Under the Curve (AUC) of Vorinostat After Single Oral Dosing | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours post-dose on Days 1 and 17

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Watanabe T, Kato H, Kobayashi Y, Yamasaki S, Morita-Hoshi Y, Yokoyama H, Morishima Y, Ricker JL, Otsuki T, Miyagi-Maesima A, Matsuno Y, Tobinai K. Potential efficacy of the oral histone deacetylase inhibitor vorinostat in a phase I trial in follicular and mantle cell lymphoma. Cancer Sci. 2010 Jan;101(1):196-200. doi: 10.1111/j.1349-7006.2009.01360.x. Epub 2009 Sep 10. PMID 19817748